CLINICAL TRIAL: NCT06045195
Title: Phase II Trial of Pembrolizumab in First-Line Treatment of Advanced-Stage Classical Hodgkin Lymphoma
Brief Title: Pembrolizumab in First-Line Treatment of Advanced-Stage Classical Hodgkin Lymphoma
Acronym: Pembro-FLASH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-4938
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
Keywords: advanced stage; first line treatment; PD-1 inhibitor
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Pembrolizumab + BrECADD
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — As induction therapy, all participants will receive one dose of single-agent pembrolizumab (P) followed by two cycles of chemo-immunotherapy consisting of pembrolizumab and BrECADD (P-BrECADD). Response to induction therapy will be measured after 1x P (PET-1) and after 1x P + 2x P-BrECADD (PET-3).
  Further systemic treatment is PET-3-guided. Complete metabolic responses will be consolidated with two further cycles of P-BrECADD while participants with a positive PET-3 will receive four further cycles of P-BrECADD. PET-positive lesions after completion of chemo-immunotherapy will be recommended for consolidating radiotherapy according to standard of care.

SUMMARY:
The primary objective of this trial is to estimate efficacy of the novel regimen. The primary endpoint is the 1-year PFS rate after treatment with one dose of pembrolizumab followed by four to six cycles of chemo-immunotherapy with P-BrECADD, and PET-guided radiotherapy as per standard of care

ELIGIBILITY:
Main Inclusion Criteria:

* age 18-60
* advanced stage classical Hodgkin Lymphoma
* no previous treatment for cHL

Main Exclusion Criteria:

* Nodular lymphocyte-predominant Hodgkin lymphoma or composite lymphoma
* Chemotherapy or radiotherapy in medical history
* Prior or concurrent disease that prevents treatment according to protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Principal Investigator — 1st Department of Medicine, Cologne University Hospital
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided